CLINICAL TRIAL: NCT05788939
Title: DOES PLANNED VISUAL EDUCATION AFFECT UNIVERSITY STUDENTS' ATTITUDES AND BELIEFS ABOUT SKIN CANCER?
Brief Title: PLANNED VISUAL EDUCATION ABOUT SKIN CANCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-186
Record Dates: First submitted 2023-03-02; First posted 2023-03-29 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Skin Neoplasm
Keywords: Health belief model; health attitudes; university students; skin cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: The sample of this cluster randomized controlled experimental study consisted of 2nd year university students (n=116) training in Faculty of Economics and Administrative Sciences (FEAS) and Hasan Ferdi Turgutlu Faculty of Technology (HFTFT) from the faculties of Manisa Celal Bayar University (MCBU) between February-Semptember 2019. Among the faculties in MCBU, simple random sampling was used to draw lots, with the first lot being assigned to FEAS as the intervention group (IG), and the second lot being assigned to HFTFT as the control group (CG) . Among seven departments in FEAS and four departments in the HFTFT, simple random sampling was used to draw lots again. The Department of Econometrics from the FEAS was assigned as the IG and Mechatronics Engineering from HFTFT was assigned as the CG.
  58 students for the CG and 58 students for the IG were recruited for the sample. Power of the study was calculated as post hoc at α=0.05 with a significance of 0.95.
Who Masked: Participant
Masking Description: Participants in the study do not know whether they are in the experimental or control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The sample of this cluster randomized controlled experimental study consisted of 2nd year university students (n=116) training in Faculty of Economics and Administrative Sciences (FEAS) and Hasan Ferdi Turgutlu Faculty of Technology (HFTFT) from the faculties of Manisa Celal Bayar University (MCBU) between February-Semptember 2019. Among the faculties in MCBU, simple random sampling was used to draw lots, with the first lot being assigned to FEAS as the intervention group (IG), and the second lot being assigned to HFTFT as the control group (CG) . Among seven departments in FEAS and four departments in the HFTFT, simple random sampling was used to draw lots again. The Department of Econometrics from the FEAS was assigned as the IG and Mechatronics Engineering from HFTFT was assigned as the CG. The planned visual education based Health Belief Model was given.
  Interventions: Other: Planned Visual Education Based on Health Belief Model
- Control group (No Intervention): No attempt was made by researcher during the study. Only data were collected. At the end of the study, the planned visual education based Health Belief Model was given and all students continued in the study were given key rings with pictures about sun protection designed by the researchers.

INTERVENTIONS:
Other: Planned Visual Education Based on Health Belief Model — The students in IG were administered the planned visual education based on Health Belief Model for a period of seven months.
  The education materials were a PowerPoint presentation, a skin cancer model, videos titled "Dear 16 years old me", "Mr. Sun", a brochure, and 3 posters.
  .
  Arms: intervention group

SUMMARY:
This study aimed to evaluate the effect of planned visual education based on the Health Belief Model on university students' attitudes and beliefs toward skin cancer. The planned visual education based in Health Belief Model has possitive effects on univestiy students' attitudes and beliefs toward skin cancer.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of planned visual education based on the Health Belief Model on university students' attitudes and beliefs toward skin cancer. Planned as a cluster-randomized controlled experimental study conducted on two groups (n=116). The study was carried out in Faculty of Economics and Administrative Sciences (FEAS) and Hasan Ferdi Turgutlu Faculty of Technology (HFTFT) from the faculties of Manisa Celal Bayar University (MCBU) between February-Semptember 2019. Among seven departments in FEAS and four departments in the HFTFT, simple random sampling was used to draw lots again. The Department of Econometrics from the FEAS was assigned as the intervation groups (n=58) and Mechatronics Engineering from HFTFT was assigned as the control group (n=58). Data were collected using The Student Introduction Form and The Health Belief Model Scale in Skin Cancer.

ELIGIBILITY:
Inclusion Criteria:

* who Registered and continuing department courses
* who agreed to participate in the study
* who had formal education
* who been second year students

Exclusion Criteria:

* Registration and absence of the student in the department courses
* Refusal to participate in the study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The Health Belief Model Scale in Skin Cancer | One months
  Developed by Dogan and Caydam (2021), the scale consists of 26 items and 5 sub-dimensions (perceived susceptibility, perceived benefit, perceived severity, perceived barriers, and self-efficacy). The HBMSSC is a five-point Likert-type scale, and each item is answered from "disagree=1" to "strongly agree=5". The total Cronbach's alpha coefficient of the scale is 0.86, and for the sub-dimensions it is 0.89; 0.79; 0.77; 0.65 and 0.86, respectively. The "perceived barriers" sub-dimension of the scale is reverse coded. The scale does not have a total score, and each sub-dimension is scored within itself. Higher "perceived susceptibility, "perceived benefit, "perceived severity", and "self-efficacy" scores indicate higher perceived susceptibility, perceived benefit, perceived severity, and self-efficacy
The Health Belief Model Scale in Skin Cancer | Three months
  Developed by Dogan and Caydam (2021), the scale consists of 26 items and 5 sub-dimensions (perceived susceptibility, perceived benefit, perceived severity, perceived barriers, and self-efficacy). The HBMSSC is a five-point Likert-type scale, and each item is answered from "disagree=1" to "strongly agree=5". The total Cronbach's alpha coefficient of the scale is 0.86, and for the sub-dimensions it is 0.89; 0.79; 0.77; 0.65 and 0.86, respectively. The "perceived barriers" sub-dimension of the scale is reverse coded. The scale does not have a total score, and each sub-dimension is scored within itself. Higher "perceived susceptibility, "perceived benefit, "perceived severity", and "self-efficacy" scores indicate higher perceived susceptibility, perceived benefit, perceived severity, and self-efficacy
The Health Belief Model Scale in Skin Cancer | Seven months
  Developed by Dogan and Caydam (2021), the scale consists of 26 items and 5 sub-dimensions (perceived susceptibility, perceived benefit, perceived severity, perceived barriers, and self-efficacy). The HBMSSC is a five-point Likert-type scale, and each item is answered from "disagree=1" to "strongly agree=5". The total Cronbach's alpha coefficient of the scale is 0.86, and for the sub-dimensions it is 0.89; 0.79; 0.77; 0.65 and 0.86, respectively. The "perceived barriers" sub-dimension of the scale is reverse coded. The scale does not have a total score, and each sub-dimension is scored within itself. Higher "perceived susceptibility, "perceived benefit, "perceived severity", and "self-efficacy" scores indicate higher perceived susceptibility, perceived benefit, perceived severity, and self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- CelalBayarU, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
ll IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: starting 6 months after publication
Access Criteria: It can be shared upon request, if the relevant ethics committee approves.

REFERENCES:
- [Result] Barbaric J, Sekerija M, Agius D, Coza D, Dimitrova N, Demetriou A, Safaei Diba C, Eser S, Gavric Z, Primic-Zakelj M, Zivkovic S, Zvolsky M, Bray F, Coebergh JW, Znaor A. Disparities in melanoma incidence and mortality in South-Eastern Europe: Increasing incidence and divergent mortality patterns. Is progress around the corner? Eur J Cancer. 2016 Mar;55:47-55. doi: 10.1016/j.ejca.2015.11.019. Epub 2016 Jan 9. PMID 26773419
- [Result] Livingstone E, Windemuth-Kieselbach C, Eigentler TK, Rompel R, Trefzer U, Nashan D, Rotterdam S, Ugurel S, Schadendorf D. A first prospective population-based analysis investigating the actual practice of melanoma diagnosis, treatment and follow-up. Eur J Cancer. 2011 Sep;47(13):1977-89. doi: 10.1016/j.ejca.2011.04.029. Epub 2011 May 24. PMID 21612915
- [Result] Birch-Johansen F, Jensen A, Mortensen L, Olesen AB, Kjaer SK. Trends in the incidence of nonmelanoma skin cancer in Denmark 1978-2007: Rapid incidence increase among young Danish women. Int J Cancer. 2010 Nov 1;127(9):2190-8. doi: 10.1002/ijc.25411. PMID 20473901
- [Result] Karagas MR, Zens MS, Li Z, Stukel TA, Perry AE, Gilbert-Diamond D, Sayarath V, Stephenson RS, Barton D, Nelson HH, Spencer SK. Early-onset basal cell carcinoma and indoor tanning: a population-based study. Pediatrics. 2014 Jul;134(1):e4-12. doi: 10.1542/peds.2013-3559. PMID 24958589
- [Result] Armstrong AW, Idriss NZ, Kim RH. Effects of video-based, online education on behavioral and knowledge outcomes in sunscreen use: a randomized controlled trial. Patient Educ Couns. 2011 May;83(2):273-7. doi: 10.1016/j.pec.2010.04.033. Epub 2010 Jun 1. PMID 20570081
- [Result] Stanton WR, Chakma B, O'Riordan DL, Eyeson-Annan M. Sun exposure and primary prevention of skin cancer for infants and young children during autumn/winter. Aust N Z J Public Health. 2000 Apr;24(2):178-84. doi: 10.1111/j.1467-842x.2000.tb00139.x. PMID 10790938
- [Result] Wesson KM, Silverberg NB. Sun protection education in the United States: what we know and what needs to be taught. Cutis. 2003 Jan;71(1):71-4, 77. PMID 12553634
- [Result] Makin JK, Warne CD, Dobbinson SJ, Wakefield MA, Hill DJ. Population and age-group trends in weekend sun protection and sunburn over two decades of the SunSmart programme in Melbourne, Australia. Br J Dermatol. 2013 Jan;168(1):154-61. doi: 10.1111/bjd.12082. PMID 23039760
- [Result] Celik S, Ilce A, Andsoy II. Knowledge and Protective Behaviors About Skin Cancer Among Nursing Students in the West Black Sea Region of Turkey. J Cancer Educ. 2018 Aug;33(4):885-892. doi: 10.1007/s13187-017-1188-5. PMID 28229313
- [Result] Balyaci OE, Kostu N, Temel AB. Training program to raise consciousness among adolescents for protection against skin cancer through performance of skin self examination. Asian Pac J Cancer Prev. 2012;13(10):5011-7. doi: 10.7314/apjcp.2012.13.10.5011. PMID 23244101
- [Result] Glanz K, Steffen AD, Schoenfeld E, Tappe KA. Randomized trial of tailored skin cancer prevention for children: the Project SCAPE family study. J Health Commun. 2013;18(11):1368-83. doi: 10.1080/10810730.2013.778361. Epub 2013 Jun 27. PMID 23806094
- [Result] Nahar VK, Ford MA, Hallam JS, Bass MA, Hutcheson A, Vice MA. Skin Cancer Knowledge, Beliefs, Self-Efficacy, and Preventative Behaviors among North Mississippi Landscapers. Dermatol Res Pract. 2013;2013:496913. doi: 10.1155/2013/496913. Epub 2013 Oct 7. PMID 24223037
- [Result] Haney MO, Bahar Z, Beser A, Arkan G, Cengiz B. Psychometric Testing of the Turkish Version of the Skin Cancer and Sun Knowledge Scale in Nursing Students. J Cancer Educ. 2018 Feb;33(1):21-28. doi: 10.1007/s13187-016-1041-2. PMID 27155664
- [Result] Khani Jeihooni A, Hidarnia A, Kaveh MH, Hajizadeh E. The effect of a prevention program based on health belief model on osteoporosis. J Res Health Sci. 2015 Winter;15(1):47-53. PMID 25821026
- [Result] Kissal A, Kartal B. Effects of Health Belief Model-Based Education on Health Beliefs and Breast Self-Examination in Nursing Students. Asia Pac J Oncol Nurs. 2019 Oct-Dec;6(4):403-410. doi: 10.4103/apjon.apjon_17_19. PMID 31572761
- [Result] Tuong W, Armstrong AW. Effect of appearance-based education compared with health-based education on sunscreen use and knowledge: a randomized controlled trial. J Am Acad Dermatol. 2014 Apr;70(4):665-669. doi: 10.1016/j.jaad.2013.12.007. Epub 2014 Feb 5. PMID 24508292
- [Result] Trinh N, Novice K, Lekakh O, Means A, Tung R. Use of a brief educational video administered by a portable video device to improve skin cancer knowledge in the outpatient transplant population. Dermatol Surg. 2014 Nov;40(11):1233-9. doi: 10.1097/DSS.0000000000000148. PMID 25310749
- [Derived] Dogan ES, Caydam OD. Effect of planned visual education on university students' attitudes and beliefs regarding skin cancer: a cluster-randomized controlled trial. Sao Paulo Med J. 2025 May 30;143(4):e2024252. doi: 10.1590/1516-3180.2024.0252.R1.14022025. eCollection 2025. PMID 40465956
- See also: World Health Organization — http://www.who.int/uv/faq/skincancer/en/index1.html
- See also: Cancer Research UK — https://www.cancerresearchuk.org/sites/default/files/sun_protection_trends_-_cruk.pdf
- Available data/document: Informed Consent Form — https://dergipark.org.tr/tr/download/article-file/820404 — Dogan ES, Caydam OD. Investigation of Studies Conducted with Health Belief Model in Skin Cancer. Izmir Democracy University Health Sciences Journal.2019; 2(2):66-75.
- Available data/document: Statistical Analysis Plan — https://saudijournals.com/media/articles/SJNHC_48_205-213.pdf — Dogan ES, Caydam OD. A Scale Development Study: Health Belief Model Scale in Skin Cancer among Turkish University Students. Saudi Journal of Nursing and Health Care. 2021; 4(8): 205- 213. https://doi.org/10.36348/sjnhc.2021.v04i08.001.